CLINICAL TRIAL: NCT02631772
Title: LIVE-C-Free: Early and Late Treatment of Hepatitis C With Sofosbuvir/Ledipasvir in Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-337-1830
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir, sofosbuvir drug combination; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Late Cohort, Arm 1 (Experimental): Ledispasvir (LDV) and Sofosbuvir (SOF) monotherapy x 12 weeks
  Interventions: Drug: Sofosbuvir/Ledipasvir x 12 weeks
- Late Cohort, Arm 2 (Active Comparator): Ledispasvir (LDV) and Sofosbuvir (SOF) +ribavirin x 12 weeks
  Interventions: Drug: Sofosbuvir/Ledipasvir + Ribavirin x 12 weeks

INTERVENTIONS:
Drug: Sofosbuvir/Ledipasvir x 12 weeks
  Other Names: Harvoni
  Arms: Late Cohort, Arm 1
Drug: Sofosbuvir/Ledipasvir + Ribavirin x 12 weeks
  Arms: Late Cohort, Arm 2

SUMMARY:
The predominant remaining questions for post-transplant treatment of Hepatitis C virus (HCV) in the DAA (direct acting anti-virals) era are whether a ribavirin-free regimen is possible and whether pre-emptive treatment is now a potential option to prevent long-term damage to the allograft.

Our aim is to provide answers to these primary questions with our multicenter, prospective, randomized, open-label intent-to-treat phase IV study

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open-label phase IV study.

Compare ledipasvir/sofosbuvir + ribavirin for 12 weeks vs ledipasvir/sofosbuvir alone for 12 weeks in patients over 90 days post-liver transplant

ELIGIBILITY:
Inclusion Criteria

1. At least 18 years of age and able to give informed consent
2. History of HCV genotype 1 or 4
3. Normal EKG
4. At least 91 days post orthotopic liver transplant
5. Screening laboratory values within defined thresholds
6. Detectable HCV RNA at screening
7. Creatinine Clearance of at least 40ml/min using the Cockcroft Gault equation
8. Negative pregnancy test for female subjects within 48 hours prior to receiving study medication
9. Use of two effective contraception methods if female of childbearing potential or sexually active male unless status post bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or vasectomy

Exclusion Criteria

1. Serious or active medical or psychiatric illness
2. History of significant or unstable cardiac disease
3. Stomach disorder that could interfere with the absorption of the study drug
4. Pregnant or nursing females or males with a pregnant female partner
5. Co-infected with Hepatits B (HBV) or HIV
6. Recipients of an allograft from a donor that was infected with HCV with an unknown genotype or non-genotype 1 or 4 unless the recipient is demonstrated to have only genotype 1 or 4 HCV replication post-transplant
7. Allergic to or intolerant of sofosbuvir, ledipasvir, or ribavirin
8. History of exposure to an Nonstructural protein (NS5A) inhibitor
9. Within 1 year of transplant AND history of Hepatocellular Carcinoma (HCC) with tumor burden outside of the Milan Criteria (See Appendix II) prior to transplant
10. Participated in a clinical study with an investigational drug or biologic within the last 30 days
11. Combined liver/kidney transplant
12. History of organ transplant other than liver
13. Childs Turcotte Pugh (CTP) B or C
14. Patients with fibrosing cholestatic hepatitis
15. Platelet count of ≤ 30 k/mm3
16. Hemoglobin < 10g/dL
17. Total bilirubin > 10mg/dL
18. Alanine aminotransferase (ALT),aspartate aminotransferase (AST), or alkaline phosphatase ≥ 10x upper limit normal
19. Serum sodium < 125mmol/L
20. Current use of any of the Prohibited Interventions (Section 5.3.2) and un-willing to discontinue use, or use of amiodarone within 6 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Late Cohort, Arm 1: LDV/SOF monotherapy x 12 weeks
  Sofosbuvir/Ledipasvir x 12 weeks
- Late Cohort, Arm 2: LDV/SOF+ribavirin x 12 weeks
  Sofosbuvir/Ledipasvir + Ribavirin x 12 weeks
Period: Overall Study
Arm/Group | Late Cohort, Arm 1 | Late Cohort, Arm 2
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Late Cohort, Arm 1 | Late Cohort, Arm 2 | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (4) | 60 (4) | 61 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 9 | 14 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Days since transplant [Mean (Standard Deviation); unit: days] | 1862 (1309) | 2611 (1998) | 2237 (1654)
Calculated MELD at Transplant [Mean (Standard Deviation); unit: units on a scale] — MELD (Model for End-Stage Liver Disease) predicts survival for patients with advanced liver disease. Scale range is as follows:
  Score Mortality Probability
  40 (71.3% mortality) 30-39 (52.6% mortality) 20-29 (19.6% mortality) 10-19 (6.0% mortality) 9 or less (1.9% mortality)
  units on a scale | 22.3 (6.4) | 24.7 (8.7) | 23.5 (7.6)
Number of patients with prior HCV Treatment [Count of Participants; unit: Participants] | 7 | 8 | 15
Number of subjects with history of depression [Count of Participants; unit: Participants] | 3 | 6 | 9
Number of subjects with history of anemia [Count of Participants; unit: Participants] | 6 | 6 | 12
Number of subjects with history of leukopenia [Count of Participants; unit: Participants] | 4 | 3 | 7
Number of subjects with history of thrombocytopenia [Count of Participants; unit: Participants] | 4 | 4 | 8
Number of subjects with history of chronic kidney disease [Count of Participants; unit: Participants] | 4 | 5 | 9
Number of subjects with history of insomnia [Count of Participants; unit: Participants] | 3 | 4 | 7
Type of HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 13 | 14 | 27
  Genotype 1b | 3 | 2 | 5
Number of subjects with resistant mutations [Count of Participants; unit: Participants]
  NS5A Resistant Mutation | 2 | 0 | 2
  NS5B Resistant Mutation | 0 | 0 | 0
Number of subjects with a previous transplant [Count of Participants; unit: Participants] | 0 | 1 | 1
Number of subjects with CMV positive serostatus [Count of Participants; unit: Participants] | 12 | 13 | 25
Percent of participants with Previous Interferon use [Number; unit: %] — Row 1 is the % of subjects who previously used interferon.
  Row 2 is the % of subjects who previously used interferon, that subsequently stopped interferon prematurely.
  %
    Previous Interferon use | 38 | 50 | 14
    Stopped interferon prematurely | 67 | 100 | 12
Number of subjects with Split Liver [Count of Participants; unit: Participants] | 1 | 2 | 3
Number of subjects with an HCV positive donor [Count of Participants; unit: Participants] | 2 | 0 | 2
Donor age [Mean (Standard Deviation); unit: years] | 36 (13) | 37 (14) | 37 (14)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy
Description: Treatment efficacy, defined as the percentage of patients achieving sustained virologic response 12 (SVR12) weeks after completing the antiviral regimen
Time Frame: 12 Weeks
Measure: Number; unit: % of participants
Arm/Group | Late Cohort, Arm 1 | Late Cohort, Arm 2
Number analyzed (Participants) | 16 | 16
% of participants | 88 | 75

2. Secondary Outcome: Number of Participants With Virologic Failure
Description: Number of participants who had a nonresponse to treatment or a relapse of disease under study.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Late Cohort, Arm 1 | Late Cohort, Arm 2
Number analyzed (Participants) | 16 | 16
Participants
  Nonresponse | 0 | 1
  Relapse | 1 | 2

3. Secondary Outcome: Hemoglobin Levels
Description: Change in hemoglobin levels over the course of the study
Time Frame: Week 4, Week 8, Week 12, Week 16
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Late Cohort, Arm 1 | Late Cohort, Arm 2
Number analyzed (Participants) | 16 | 16
g/dL
  Hemoglobin levels at Week 4 | 13.1 (2.3) | 12.9 (1.5)
  Hemoglobin levels at Week 8 | 13.3 (1.7) | 11.2 (1.7)
  Hemoglobin levels at Week 12 | 13.7 (1.9) | 12.0 (2.3)
  Hemoglobin levels at Week 16 | 13.6 (1.9) | 13.1 (1.9)

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Late Cohort, Arm 1 | Late Cohort, Arm 2
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 4/16 | 12/16
Other Adverse Events (participants affected / at risk) | 11/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Late Cohort, Arm 1 (N=16) | Late Cohort, Arm 2 (N=16)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fractured hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastrointestinal Syndrom (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Intermittent Complete heart block (Cardiac disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Recurrent falls when walking (General disorders) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
COPD (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Late Cohort, Arm 1 (N=16) | Late Cohort, Arm 2 (N=16)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 11 (11)
Fatigue (General disorders) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Increased creatinine (Renal and urinary disorders) | 2 (2) | 7 (7)
Insomnia (General disorders) | 0 (0) | 2 (2)
headache (General disorders) | 2 (2) | 2 (2)
Increased liver function tests (Hepatobiliary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT02631772/Prot_SAP_000.pdf